CLINICAL TRIAL: NCT03360799
Title: A Comparison of the Attitudes About Legalization of Marijuana Use for Medical Purposes by Cancer Patients in Two Cancer Centers Located in a Legalized and a Non-Legalized State
Brief Title: Questionnaires in Assessing Attitudes About Legalization of Marijuana Use in Participants With Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0568; NCI-2018-01026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0568 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire): Participants complete 5 questionnaires.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies attitudes about legalization of marijuana use in participants with cancer. Questionnaires may help doctors to learn about and compare the attitudes that patients in non-legalized and legalized states have towards the legalization of medical marijuana.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the proportion of cancer patients' who have a positive attitude about legalizing marijuana for medical purposes between those in a legalized versus (vs.) a non-legalized state.

SECONDARY OBJECTIVES:

I. To evaluate the association of cancer patients' belief in the usefulness of medical marijuana in their state of residency (Texas versus Arizona).

II. To examine the association of demographic, physical and psychosocial characteristics of patients and their perception of medical marijuana.

III. To examine the preference of patients for treatment of pain, anxiety and depression between medical marijuana vs. opioids, anti-anxiety and anti-depressant medications.

IV. To examine the association of media to perception of use of medical marijuana.

V. To evaluate the association of cancer patients' attitude about legalizing marijuana for medical purposes vs. recreational purposes.

VI. To examine the association of patients who have used marijuana for certain medical conditions/symptoms and their belief of how it has affected that condition/symptom.

VII. To compare demographic, physical and psychosocial characteristics of patients who have used marijuana for medical purposes.

VIII. To compare demographic, physical and psychosocial characteristics of patients who have used marijuana for non-medical purposes. IX. To compare demographic, physical and psychosocial characteristics of patients who believe marijuana is useful for medical reasons.

OUTLINE:

Participants complete 5 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients (inpatient or outpatient) seen by the Palliative Care team at Banner MD Anderson or UT MD Anderson
* Patients able to speak and read English
* Patients enrolled in each site must be a resident of the state where that site is located (e.g. if a patient is enrolled at UT MD Anderson Cancer Center [MDACC], they should be resident of the state of Texas)
* Patients should have a cancer diagnosis

Exclusion Criteria:

* Patients who are not able to speak or read English
* Altered mental status as determined by the interviewer based on the ability to understand the nature of the study and consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with cancer seen by the Palliative Care team at Banner MD Anderson or University of Texas (UT) MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Positive attitude regarding the legalization of medical marijuana for medical purposes | Up to 1 year
  Will be defined as answering "Completely Agree" or "Slightly Agree" to the question 1 in Marijuana Survey for Patients. The number of subjects with positive attitude towards legalizing medical marijuana will be compared between patients from Texas and Arizona States using one-sided Fisher's exact test or chi-squared test, whichever appropriate. A logistic model will be used to assess the effect of state of residency, adjusting for other covariates such as gender, age, race, etc. Will employ inverse probability of state weighting using the propensity score on all patients to estimate the difference in attitudes of marijuana use between the states. In the weighted sample, will also compute the standardized differences to evaluate the balance of baseline covariates between the two states. The propensity score model may be adjusted to further minimize some of the residual difference in the distribution of the baseline covariates between the two states.

SECONDARY OUTCOMES:
Participants' belief in the usefulness of medical marijuana between those who are residents of Texas versus Arizona | Up to 1 year
  The proportion of patients with positive belief will be reported with a 95% confidence interval. Fisher's exact test will be applied to compare the proportion between residents of two states.
Perception of medical marijuana | Up to 1 year
  Will evaluate the association of demographical, physical, and psychosocial characteristics of patients and their perception of medical marijuana. In order to address this objective, all the specified characteristics will be summarized by descriptive statistics based on patients' perception of medical marijuana (positive or negative attitude); chi-square (or Fisher's exact) test and Wilcoxon rank sum test may be applied to test the associations for categorical and continuous variables, respectively. Logistic regression model may be utilized to evaluate the association of patients' characteristics with their perception of medical marijuana. Summarized reports of all other questions regarding the preference of patients for treatment of pain, anxiety and depression between medical marijuana versus opioids, anti-anxiety, anti-depressant medications, as well as the perception of impact of media on patient's preference in the Marijuana Survey for Patients will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberson C Tanco, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org